CLINICAL TRIAL: NCT06603532
Title: Effect of Low-Load Blood Flow Restricted Training on Volitional Activation of Knee Extensor Muscles in Subjects with Knee Joint Impairment
Brief Title: Effect of LL-BFRE Training on Volitional Muscle Activation in Subjects with Knee Joint Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana (Other)
Collaborators: University Medical Centre Ljubljana (Other); University of Primorska (Other)
Responsible Party: Principal Investigator, Alan Kacin, Head of Laboratory, University of Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0120-496-2018-8; P3-0043 (Other Grant/Funding Number: Slovenian Research and Innovation Agency); 20190041; 20200063 (Other Grant/Funding Number: University Clinical Center Ljubljana)
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Arthrogenic Muscle Inhibition; Knee Injuries; Knee Surgery
Keywords: arthrogenic muscle inhibition; knee injury; level of volunaty muscle activation; blood flow restriction resistance exercise; controlled clinical trial
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Intervention Model Description: prospective, single-center, double-blinded, quasi-randomized controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- low-load blood flow restriction (BFR) resistance training (Experimental): Group of patients that performed the experimental exercise training against low mechanical resistance (workload) with blood flow restriction (BFR) in the active thigh muscles.
  Interventions: Other: low-load blood flow restriction (BFR) training
- low-load resistance training (Sham Comparator): Group of patients that performed exercise training against low mechanical resistance (workload) with sham blood flow restriction (SHAM-BFR) in the active thigh muscles.
  Interventions: Other: low-load resistance training

INTERVENTIONS:
Other: low-load blood flow restriction (BFR) training — The training program lasted four weeks with three training sessions per week, for a total of 12 training sessions. Participants in the BFR group exercised with blood flow restriction caused by an inflatable cuff placed on the proximal part of the thigh and inflated to 120-140 mmHg. Subjects trained against the maximum mechanical resistance they could overcome thirty times (30 repetitions maximum; 30 RM). All training sessions were performed under the supervision of a physiotherapist and included leg press and knee extension exercises.
  Arms: low-load blood flow restriction (BFR) resistance training
Other: low-load resistance training — The training program lasted four weeks with three training sessions per week, for a total of 12 training sessions. Participants in SHAM-BFR group performed an identical exercise protocol as experimental (BFR) group, while having thigh cuff inflated to only 20 mmHg, which did not affect normal muscle blood flow. Subjects trained against the maximum mechanical resistance they could overcome thirty times (30 repetitions maximum; 30 RM). All training sessions were performed under the supervision of a physiotherapist and included leg press and knee extension exercises.
  Arms: low-load resistance training

SUMMARY:
The aim of this study was to investigate whether 4 weeks of exercise training against low mechanical resistance in combination with partial blood flow restriction has an additional therapeutic effect on the patients' ability to activate the knee extensor muscle. Patients with chronic deficits in muscle strength due to knee injuries or surgery on one leg were invited to participate in this study on a completely voluntary basis.

DETAILED DESCRIPTION:
The effects of low-load exercise with blood flow restriction (BFR) on the ability to voluntarily activate skeletal muscle in people with joint injuries are poorly understood. The aim of our study was to investigate the effects of low-load BFR training on the level of voluntary activation (AL) of the quadriceps femoris muscle assessed using the interpolated twitch technique in people with different knee joint injuries. Thirty-three orthopedic patients assigned to either the BFR group or the SHAM-BFR group participated in the study. Over a period of four weeks, the participants completed 12 training sessions of unilateral knee extension and leg press at 30 RM. The BFR group trained with a pneumatic cuff-induced blood flow restriction (pressure = 120-140 mmHg), while the SHAM-BFR group trained with a sham blood flow restriction (pressure = 20 mmHg) that did not interfere with normal muscle perfusion. The assessment of knee muscle capacity and function consisted of dynamometric measurements of maximal isometric strength and endurance of the knee extensor muscles, level of voluntary muscle activation, surface electromiography, pain intensity and assessment of perceived exertion. All tests and measurements were performed twice, once before the intervention (baseline) and once at the end of the 4-week training period (POST).

ELIGIBILITY:
Inclusion Criteria:

* no systemic illness,
* no history of injuries to the contralateral knee,
* pain intensity during exercise ≤ 2 on numeric pain rating scale (0-10).

Exclusion Criteria:

* neuromuscular impairments,
* spine or other lower limb injuries,
* presence or history of any vascular diseases or deep vein thrombosis
* pain intensity during exercise ≥ 3 on numeric pain rating scale (0-10).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Quadriceps muscle isometric strength | Baseline and 4 weeks (post intervention)
  The measurement of the torque of the maximum volitional isometric contraction (MVIC) of the quadriceps femoris (QF) was performed on an isometric knee joint dynamometer. The test subject was seated, the hip joint was flexed to 85° and the lever arm was locked at 60° knee flexion. After warming up, the subject was instructed to perform the MVIC for 3-5 seconds with arms crossed over the chest, with no upper body movements allowed. Three consecutive MVICs were performed with each leg, separated by a 30-second rest period. The experimenter gave the subjects strong verbal encouragement during the tests. The highest average 1-second torque (Nm) of the three trials was considered relevant and used for further analysis.
Maximal voluntary activation level of quadriceps muscle | Baseline and 4 weeks (post intervention)
  The degree of QF maximal voluntary activation (VAmax) was calculated as the ratio between the highest interpolated twitch contraction torque achieved during MVIC and the highest muscle twitch torque at rest measured during the first 10-second recovery period of after MVIC. The value is expressed as a percentage (%).
Quadriceps muscle isometric endurance | Baseline and 4 weeks (post intervention)
  The test of QF isometric endurance was performed on an isometric knee joint dynamometer. The test subject was seated with the hip joint flexed to 85° and the lever arm locked at 60° knee flexion. After warming up, the test subject was instructed to attain 60% MVIC torque displayed on a computer screen and to maintain this until voluntary failure. The experimenter gave the subjects strong verbal encouragement during the test. QF muscle endurance was measured in seconds (s).
Voluntary activation level of quadriceps muscle during isometric endurance test | Baseline and 4 weeks (post intervention)
  The degree of QF voluntary activation was evaluated in 10-s intervals during the isometric endurance test (VAendur). It was calculated as the ratio between the twitch torque attained in a given time interval and the highest muscle twitch torque at rest measured during the 20-second recovery period after the test. The value was expressed as a percentage (%).
Surface EMG amplitude of quadriceps muscle during isometric endurance test | Baseline and 4 weeks (post intervention)
  The change in activation of v. medialis, v. lateralis and rectus f. muscles was measured using surface EMG during the isometric endurance test. The electrodes were positioned according to the SENIAM standards (Hermens et al., 2000) to avoid overlapping of the innervation zones and cross-talk between the muscles. EMG activity was amplified using a four-channel monitoring device with a sampling rate of 1000 Hz, an input impedance of 2MΏ and a bandwidth of 1-500 Hz. Smoothing the root mean square (RMS) of the filtered signal with a time window of 3000 ms was used to quantify the EMG amplitude (mV). The RMS EMG during the endurance test was expressed as percentage of the highest value attained during MVIC (% RMS EMG max).

SECONDARY OUTCOMES:
knee and muscle pain | during each training session, 3-times per week, for 4 weeks
  The intensity of pain at rest and at the end of each exercise repetition was rated using a numerical pain scale (NPRS) from 0-10, with 0 is the absence of pain and 10 is the worst pain imaginable.
ratings of perceived exertion | during each training session, 3-times per week, for 4 weeks
  Ratings of perceived exertion (RPE) were assessed at the end of each exercise set using the Borg 10 category-ratio scale, with 0 is no effort and 10 is an extreme physical effort.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Kacin, PhD, PT, Prof, Principal Investigator — University of Ljubljana, Faculty of Health Studies
Locations (2):
- Slovenia (2):
  - University of Primorska, Faculty of Health Sciences, Izola
  - University of Ljubljana, Faculty of Health Sciences, Ljubljana

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD in anonymized form.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: No limit.
Access Criteria: All IPD will be shared upon reasoned request for the purpose of further scientific analysis (i.e. systematic reviews, meta-analyzes, etc.). A proposal describing the planned analyzes must be submitted in writing to the principal investigator, Dr. Alan Kacin, by email to alan.kacin@zf.uni-lj.si.